

# **Trial Statistical Analysis Plan**

c03413910-02

**BI Trial No.:** 1289.27

Title: Randomised, parallel-group, double-blind study of systemic and

ocular safety and pharmacokinetics of BI 409306 in patients with schizophrenia, Alzheimer's disease, and age-comparable healthy

volunteers

**Including Protocol Amendment 3** 

1289.27-revised-protocol-03 [c02218444-07]

Investigational

**Product:** 

BI 409306

Responsible trial statistician:

TEL: FAX:

Date of statistical

08 August 2017 REVISED

analysis plan:

Version: Revised

Page 1 of 35

**Proprietary confidential information** 

 $\hbox{@ 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.}$ 

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

#### **TABLE OF CONTENTS** 1.

| $\mathbf{T}$ | ITLE P | AGE | 1 |
|---|---|---|---|
| 1. | T | ABLE OF CONTENTS | 2 |
| L | | TABLES | |
| 2. | | IST OF ABBREVIATIONS | |
| <br>3. | | NTRODUCTION | |
| ۶.<br>4. | | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY. | |
| 5. | | NDPOINTS PRIMARY ENDPOINT | |
| | 5.1<br>5.2 | SECONDARY ENDPOINTS | |
| | 5.2.1 | | |
| | 3.2.1 | (Other) Secondary Chaponits | |
| 6. | G | GENERAL ANALYSIS DEFINITIONS | 12 |
| | 6.1 | TREATMENTS | |
| | 6.2 | IMPORTANT PROTOCOL VIOLATIONS | |
| | 6.3 | SUBJECTS SETS ANALYSED | 16 |
| | | , | 16 |
| | 6.5 | POOLING OF CENTRES | |
| | 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| | <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| 7. | P | LANNED ANALYSIS | |
| | <b>7.1</b> | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| | 7.2 | CONCOMITANT DISEASES AND MEDICATION | |
| | 7.3 | TREATMENT COMPLIANCE | |
| | 7.4 | PRIMARY ENDPOINT | |
| | 7.5 | SECONDARY AND FURTHER ENDPOINTS | |
| | 7.5.1<br>7.5.2 | | |
| | 1.5.2 | (Other) Secondary endpoints | |
| | 7.7 | EXTENT OF EXPOSURE | |
| | 7.8 | SAFETY ANALYSIS | |
| | 7.8.1 | Adverse events | |
| | 7.8.2 | | |
| | 7.8.3 | · | |
| | 7.8.4 | ECG | |
| | 7.8.5 | Others | 22 |
| 8. | R | EFERENCES | 23 |
| | | ••••• | 24 |
| | | •••••• | |
| | | | 27 |

# **Boehringer Ingelheim**

| | | 27 |
|----|---------------|----|
| | | 28 |
| | | 33 |
| 10 | HISTORY TARLE | 35 |

### LIST OF TABLES

| Table 6.1: 1 | Treatment regimens / study intervals | 13 |
|--------------|-------------------------------------------------------|----|
| Table 6.1: 2 | Adverse events analysing treatment: 'Active + 7 days' | 14 |
| Table 6.2: 1 | Important protocol violations | 15 |
| Table 6.3: 1 | Subject sets analysed | 16 |
| | | 24 |
| | | 28 |
| | | 29 |

#### LIST OF ABBREVIATIONS 2.

| Term | Definition / description |
|---|---|
| AD | Alzheimer's Disease / Alzheimer's Dementia |
| AE | Adverse Event |
| AESI | Adverse Events of Special Interest |
| ATC | Anatomical Therapeutic Chemical |
| AUC | Area under the Curve |
| BDS | Biostatistics & Data Sciences |
| BI | Boehringer Ingelheim |
| BP | Blood Pressure |
| BPM | Beats Per Minute |
| BRPM | Blinded report planning meeting |
| CARE | Clinical data Analysis and Reporting Environment |
| CDR | Clinical Data Repository |
| CIAS | Cognitive Impairment Associated with Schizophrenia |
| $C_{max,ss}$ | Maximum concentration of the analyte in plasma at steady state |
| conc. | concentration |
| CPPL | Clinical Pharmacology Program Leadership |
| CRF | Case Report Form |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CYP | Cytochrome P450 |
| eCFR | electronic Case Report Form |
| ECG | Electrocardiogram |
| LCG | Licenocardiogram |
| EMEA | European Agency for the Evaluation of Medicinal Products |
| ЕоТ | End-of-Text |
| EOT | End of Trial |
| EX | Exclusion criteria from CTP |
| geom. | geometric |
| HR | Heart Rate |
| HV | Healthy Volunteer(s) |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| IDC | International Development Committee |
| IMC | International Medical Committee |
| IN | Inclusion criteria from CTP |
| IPV | Important Protocol Violation |
| | • |
| iPROG | independent Programmer |

| Term | Definition / description |
|---|---|
| iSTAT | independent Statistician |
| MedDRA | Medical Dictionary for Regulatory Activities |
| N | Number of subjects |
| O*C | Oracle Clinical |
| PAC | Premature Atrial Complexes |
| PCPK | Project Clinical PharmacoKineticist |
| PDM | Project Data Manager |
| PK | Pharmacokinetics |
| PKA | Pharmacokinetics Analyst |
| PKProg | PK Programmer |
| PKS | Pharmacokinetic Set |
| PMW | Project Medical Writer |
| PPROG | Project Programmer |
| PR | Pulse Rate |
| PSTAT | Project Statistician |
| PVC | Premature Ventricular Contraction |
| QD | quaque die (once a day) |
| QRS | Combination of Q, R and S waves |
| RAGe | Report Appendix Generator |
| R on T | refers to the R wave of the premature beat being so premature that it |
| It on 1 | coincides with the T wave of the previous beat |
| RR | ECG interval from the peak of the R wave to the peak of the subsequent |
| KK | R wave |
| SAS | Statistical Analysis System (SAS® System, SAS Institute Inc., Cary, |
| SAS | North Carolina) |
| SD | Standard Deviation |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SOC | · |
| STATANA | System Organ Class<br>Statistical analysis |
| SVT | Supraventricular |
| | 1 |
| TA | Therapeutic Area |
| TAC | Therapeutic Area Committee |
| TAH | Therapeutic Area Head |
| TALT | Therapeutic Area Leadership Team |
| TCM | Trial Clinical Monitor |
| TCPK | Trial Clinical PharmacoKineticist |
| TCPKa | Trial Clinical PharmacoKinetics Analyst |
| TDM | Trial Data Manager |
| $t_{\text{max,ss}}$ | time from dosing to maximum measured concentration of the analyte in |
| m) (T) | plasma at steady-state |
| TME | Team Member |
| TMM | Team Member Medicine |

| Term | Definition / description |
|-------|---------------------------------|
| TMW | Trial Medical Writer |
| TProg | Trial Programmer |
| TS | Treated Set |
| TSAP | Trial Statistical Analysis Plan |
| TSTAT | Trial Statistician |
| V | Visit |
| VT | Ventricular |
| WHO | World Health Organization |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 3. INTRODUCTION

TSAP for BI Trial No: 1289.27

As per ICH E9, the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

SAS® Version 9.4 or higher will be used for all analyses.

#### CHANGES IN THE PLANNED ANALYSIS OF THE STUDY 4.

There are no changes to the planned analysis described in the CTP.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 5. ENDPOINTS

This trial is designed to evaluate the ocular and systemic safety and pharmacokinetics during a 14-day treatment period in patients with schizophrenia, Alzheimer's disease, and age-comparable healthy volunteers treated with oral film-coated tablet of BI 409306 25 or 100 mg.

### 5.1 PRIMARY ENDPOINT

The primary endpoint is:

• The number (%) of subjects with AEs, coded to the MedDRA-SOC 'Eye disorders', as determined by the investigator at End of Trial

### 5.2 SECONDARY ENDPOINTS

### 5.2.1 (Other) Secondary endpoints

Secondary endpoints include:

• The number (%) of subjects with drug-related AEs as determined by the investigator at End of Trial

The following two pharmacokinetic parameters of BI 409306 are also secondary endpoints:

- C<sub>max,ss</sub> maximum measured concentration of the analyte in plasma at steady-state
- t<sub>max,ss</sub> time from dosing to maximum measured concentration of the analyte in plasma at steady-state.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

For basic study information on treatments to be administered, assignment of subjects to dose group, and selection of doses, see CTP, Section 4.

The two dose levels for this trial are described as following:

| Long label | Short label |
|---------------------|-------------|
| BI 409306 25 mg QD | BI 25mg QD |
| BI 409306 100 mg QD | BI 100mg QD |

The populations for this trial are described as: Alzheimer's Dementia (AD), cognitive impairment associated with schizophrenia (CIAS), and healthy volunteers (HV). Populations will be determined using 'Group under which subject is entering trial' captured on the demographics page at visit 1. For some displays, HV will be split into two groups: healthy volunteers comparable in age to AD subjects (HV\_AD) and healthy volunteers comparable in age to CIAS subjects (HV\_CIAS). HV\_CIAS are all HV subjects from site . HV\_AD are all HV subjects from sites . and .

| Short label unblinded | Interval<br>blinded | Sort order | CRF field |
|---|---|---|---|
| AD | AD | 01 | |
| CIAS | CIAS | 03 | |
| HV | HV | 05 | Group under which subject is entering trial |
| HV_AD | HV_AD | 02 | Group under which subject is entering that |
| HV_CIAS | HV_CIAS | 04 | |
| Total | Total | 06 | |

The following column headers will be used in the CTR displays.

The 7-column display shows population by dose and Total.

| AD | | CIAS | | HV | | |
|---|---|---|---|---|---|---|
| BI 25mg QD | BI 100mg QD | BI 25mg QD | BI 100mg QD | BI 25mg QD | BI 100mg QD | Total |

The 4-column display shows populations and Total

| | 1 1 | | |
|----|------|----|-------|
| AD | CIAS | HV | Total |

Tables displaying HV split into two groups will have the following layouts:

| 1 7 0 | 1 0 1 | |
|-------|---------|-------|
| AD | HV_AD | Total |
| and | | |
| CIAS | HV_CIAS | Total |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The 3-column display shows dose and Total

| BI 25mg QD BI 100mg QD | Total |
|------------------------|-------|
|------------------------|-------|

The following treatment phase definitions will be applied to the analyses of data except adverse events:

The **screening phase** will be defined as the time from informed consent to the date of Visit 2 (sites and ) or Visit 2 minus 1 day (site ).

The **baseline phase** will be defined as the date of Visit 2 (sites and ) or Visit 2 minus 1 day (site ) to (one minute before) the first administration of trial medication.

The **on-treatment phase** will be defined as the time from first administration of trial medication to last visit with trial medication intake.

The **post-treatment phase** will be defined as starting on the day after the last visit with drug intake to end of trial visit.

The **post-study phase** will be defined as starting from 0:00 a.m. on the day after the end of trial visit onwards.

Table 6.1: 1 Treatment regimens / study intervals

| Short label unblinded | Interval<br>blinded | Sort order+ | Start date (CRF) | Start time<br>(CRF/derived) |
|---|---|---|---|---|
| Screening | Screening | 01 | V1, Date of informed consent | 00:00 |
| Baseline For site * For sites & # | Baseline Baseline | 02 | V2, Date of visit – 1 day V2, Date of visit | 00:00 |
| 25 mg QD or<br>100 mg QD | Treat | 03 | V3, Date of study drug intake | V3, Time of study drug intake |
| Post-treatment | Post-treat | 04 | From EOT page, Date of last administration of trial drug + 1 day | V16, Time of study drug intake |
| Post-study | Post-study | 05 | EOT visit, Date of visit + 1 day | 00:00 |

<sup>+</sup> The sort order refers to the unblinded regimens.

<sup>\*</sup> Site (subjects ) is using the date of randomization to populate the visit 2 date (Using the CTP flowchart notation, this is Day -1). The date that the subject checked into the site is Day -2. This will be the start of the Baseline period and will be derived by subtracting one day from the visit 2 date.
# Sites & (subjects ) are not admitting any patients for in-patient stays. At these sites, the date of randomization is the visit 2 date and is the start of the Baseline period.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.1: 2 Adverse events analysing treatment: 'Active + 7 days'

| Label | Sort order | Start date (CRF) | Stop date |
|---|---|---|---|
| Screening | 01 | V1, Date of informed consent | V2, Date of visit 2 – 1 day* or V2, Date of visit 2 <sup>#</sup> |
| Baseline | | V2, Date of visit 2 – 1 day* or V2, Date of visit 2 <sup>#</sup> | V3, Date of study drug intake |
| Treatment | 02 | V3, Date of study drug intake | From EOT page, Date of last administration of trial drug + 1 day + 7 days |
| Post-treatment | 03 | From EOT page, Date of last administration of trial drug + 1 day + 7 days | EOT visit, Date of visit + 1 day |
| Post-study | 04 | EOT visit, Date of visit + 1 day | Date of data base lock |

<sup>\*</sup>Site

The treatment phase definitions for adverse events analyses are described above in Table 6.1: 2. All adverse events occurring from informed consent until the day before visit 2 (site ) or the day of visit 2 (sites & ) will be assigned to "screening". All adverse events occurring the day before visit 2 (site ) or the day of visit 2 (sites & ) until first dose of study drug will be assigned to "baseline". All adverse events occurring between first dose of study drug until 7 days (inclusive) after last treatment administration will be assigned to "treatment". Adverse events occurring after this period and prior to end-of-trial will be assigned to "post-treatment". Adverse events occurring after end-of-trial will be considered "post-study".

### 6.2 IMPORTANT PROTOCOL VIOLATIONS

The following table defines the different categories of important protocol violations (IPVs). The final column describes which IPVs will be used to exclude subjects from the different subject analysis sets.

<sup>\*</sup>Sites &

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.2: 1 Important protocol violations

| Category/<br>Code | | Description | Example/Comment | Potentially excluded from |
|---|---|---|---|---|
| A | | Entrance criteria not met | | |
| | A1 | Inclusion criteria not met | | |
| | A1.1 | Diagnoses of schizophrenia not | IPV if any of the clinical features defining | None |
| | | established | the population (IN1) are not met. | |
| | A1.2 | Diagnosis of AD not established | IPV if any of the clinical features defining | None |
| | | | the population (IN1) are not met | |
| | A2 | Exclusion criteria met | | |
| | A2.1 | Presence of active ocular conditions | Any of EX1-EX4 are met. | None |
| | A2.2 | Suicidal ideation or behavior | Any of EX13-EX14 | None |
| | A2.3 | Other clinically relevant baseline | Any of EX12, 15, 17-22, 24-26, 28 | None |
| | | conditions | | |
| В | | Informed consent | | |
| | B1 | Informed consent not available/not | Informed consent date missing; no | All |
| | | done | signature on ICF | |
| | <b>B2</b> | Informed consent too late | Informed consent date <actual consent<="" td=""><td>None</td></actual> | None |
| | | | date> was after Visit 1 date < Visit 1 date> | |
| $\mathbf{C}$ | | Trial medication and | | |
| | | randomisation | | |
| | C1 | Incorrect trial medication kit | Medication (kit) number assigned is not | None |
| | | assigned | from the correct group (AD, CIAS etc.). | |
| | | | OR Medication number was not assigned | |
| | | | in sequential order (as subjects were | |
| | | | randomized). | |
| | C2 | Incorrect trial medication administered | | |
| | C2.1 | Incorrect trial medication | Trial medication administered on any of | None |
| | | administered on any of days 2-13. | days 2-13 was not from the medication kit | |
| | | | assigned to subject. | |
| | C2.2 | Incorrect trial medication | Subject was administered medication from | PKS |
| | | administered on PK day 1 or 14. | kit assigned to another subject on days 1 or | |
| | | | 14 (PK visit) | |
| | <b>C3</b> | Medication code broken | Medication code broken inappropriately - | None |
| | | inappropriately | reason for medication code break | |
| | | | <reason></reason> | |
| D | | Concomitant medication | | |
| | D1 | Prohibited medication use 3 days | Use of St. Johns wort, Carbamazepine, | None |
| | | prior to Day 1 and/or Day 14. | extracts from Gingko, artemisinin, | |
| | | | enzalutamide, efavirenz, lopinavir, | |
| | | | ritonavir, tipranavir, & rifampicin. | |
| F | | Incorrect timing | | |
| | F1 | Peak exposure visual procedures | Visual procedures were not completed | None |
| | | performed outside time range. | during estimated peak exposure time range | |
| | | | (between Day 5 and Day 10 (except Day | |
| | | | 7), 20-90 minutes after dosing). | |
| Z | | Other | | |
| | <b>Z</b> 3 | Other protocol violations affecting | | None |
| | | safety only | | |

PKS: PK set

**Note**: Missing visits, evaluations, and tests will be considered missing data, not protocol deviations. All final decisions as to whether any deviation is relevant will be taken at the BRPM.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 6.3 SUBJECTS SETS ANALYSED

#### • Randomised set:

This subject set includes all randomised subjects, whether treated or not.

### • Treated set (TS):

This subject set includes all subjects who were documented to have been administered at least one dose of investigational treatment.

### • Pharmacokinetic set (PKS):

This subject set includes all subjects in the treated set who provide at least one evaluable observation for at least one PK endpoint without important protocol violations relevant to the evaluation of PK.

Table 6.3: 1 Subject sets analysed

| | Subject set | |
|---|---|---|
| Class of endpoint | Treated set | Pharmacokinetics set |
| Primary endpoint | X | |
| (other) Secondary and further endpoints | X | X |
| Safety endpoints | X | |
| Demographic/baseline endpoints | X | |
| Pharmacokinetics analysis | | X |

In addition, the population group is defined as Alzheimer's Dementia group, schizophrenia group and healthy volunteer group. The ophthalmological assessment will be done by population group.

### 6.5 POOLING OF CENTRES

This section is not applicable.

### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

With respect to safety evaluations, it is not planned to impute missing values other than AE start dates and times. Missing or incomplete AE dates are imputed according to BI standards (see "Handling of missing and incomplete AE dates"). (1)

For handling of missing data in PK evaluation, refer to CTP Appendix Section 10.1.2 and 029-DCP-102. (2)

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Unless otherwise specified, the baseline is the last available measurement before the first trial medication intake. For laboratory data that were repeatedly measured, baseline is defined to be the last available measurement before the first trial medication intake.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7. PLANNED ANALYSIS

No statistical hypothesis testing is planned. Variables will be evaluated by descriptive statistical methods in this trial.

For End-Of-Text (EoT) tables, the set of summary statistics is: N / Mean / SD / Min / Median / Max.

For displays that are provided for endpoints with some extreme data, median, quartiles and percentiles should be preferred to mean, standard deviation, minimum and maximum

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group (unless otherwise specified, all subjects in the respective subject set whether they have non-missing values or not). Percentages will be rounded to one decimal place. The category missing will be displayed only if there are actually missing values.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report, based on the TS. The following variables will be displayed: gender, age, race, ethnicity, height, weight, body mass index, smoking and alcohol status.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Only descriptive statistics are planned for this section of the report. The concomitant disease will be summarized by MedDRA primary system organ class and preferred term. The concomitant medications taken at baseline and those while on treatment will be coded using the WHO Drug coding dictionary. Concomitant medications will be summarized by WHO Drug ATC coding.

#### 7.3 TREATMENT COMPLIANCE

On each treatment day, study drug is administered to the subject at the study centre or at the ophthalmology site. Date and time of study drug intake is documented on day 1-14 of the treatment interval.

#### 7.4 PRIMARY ENDPOINT

Ocular adverse events will be those events coded to the SOC 'Eye disorders' determined by the investigator at end of trial. The assessment of ocular adverse events will be done on treated set. Ocular adverse events analyses will be performed in accordance with BI standards, essentially, tabulations of frequencies will be displayed. Refer to Section 7.8.1 for a description of the analysis of adverse events.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7.5 SECONDARY AND FURTHER ENDPOINTS

### 7.5.1 Key secondary endpoints

This section is not applicable as no key secondary endpoint has been specified in the protocol.

### 7.5.2 (Other) Secondary endpoints

Summary of drug-related AEs as determined by the investigator at end of trial will be performed in accordance with BI standards, essentially, tabulations of frequencies will be displayed. Refer to Section 7.8.1 for a description of the analysis of adverse events.

The analysis of standard PK parameters,  $C_{max,ss}$  and  $t_{max,ss}$ , will be performed as described in CTP Section 7.3.5 and also according to 029-DCG-103 ( $\underline{3}$ ). Descriptive analyses are planned.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.7 EXTENT OF EXPOSURE

Extent of exposure will be summarized by treatment group using descriptive statistics for days of exposure as well as number (percent) of patients whose total exposure falls in the following categories:

1 day, 2 days, 3 days, 4 days, etc. until 14 days, and >=15 days

Exposure to treatment will be calculated as study drug stop date minus study drug start date plus 1. Total exposure will summarize exposure to both doses.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the treated set.

### 7.8.1 Adverse events

The analyses of adverse events (AEs) will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and NOT on the number of AEs. AEs will be coded using the Medical Dictionary for Drug Regulatory Affairs (MedDRA).

For analysis, multiple AE occurrence data on the CRF will be collapsed into an AE provided that all of the following applies:

- All AE attributes are identical (LLT, intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AE of special interest).
- The occurrences were time-overlapping or time-adjacent (time-adjacency of 2 occurrences is given if the second occurrence started ≤ 24 hours from the end of the first occurrence).

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For further details on summarization of AE data, please refer to the guideline 'Handling and summarization of adverse event data for clinical trial reports and integrated summaries' (4) [001-MCG-156].

The relationship of an AE to the study drugs treatments will be assessed by the investigator.

The analysis of AEs will be based on the concept of treatment-emergent AEs. That means that all AEs occurring between first study drug intake till 7 days (inclusive) after last study drug intake will be considered "treatment-emergent" and be assigned to the randomised treatment. AEs occurring before first study drug intake will be assigned to 'screening' or 'baseline'; AEs occurring after last study drug intake + 7 days till end-of-trial visit will be assigned to 'post-treatment' (for listings only). AEs occurring after the end-of-trial visit will be assigned to 'post-study' (for listings only). For details on the treatment definition, see Section 6.1.

According to ICH E3 (5), AEs classified as 'other significant' needs to be reported and will include those non-serious and non-significant adverse events with

- (i) 'action taken = discontinuation' or 'action taken = reduced', or
- (ii) marked haematological and other lab abnormalities or lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at a Medical Quality Review Meeting.

Overall summaries of adverse events will be presented to summarise any AEs, severe AEs, drug-related AEs, AEs leading to treatment discontinuation, serious AEs, drug-related serious AEs, and AEs leading to death.

The frequency of subjects with adverse events will be summarised by treatment, primary system organ class and preferred term. Separate tables will be provided for subjects with other significant adverse events according to ICH E3 (5), for subjects with adverse events of special interest (AESI) and for subjects with serious adverse events. The AESI are described in Section 5.2.2.1 of the CTP. There is a field on the eCRF for the site to designate that an AE is an AESI. This variable will be used to identify the AESI.

The system organ classes will be sorted alphabetically, preferred terms will be sorted by frequency (within system organ class).

#### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards (6).

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7.8.3 Vital signs

Descriptive statistics of vital signs (BP and PR) observed values and change from baseline will be provided for both supine and standing positions separately. Orthostatic BP and PR will also be summarized descriptively. Orthostatic changes in BP are flagged for falls in systolic blood pressure of at least 20 mm Hg or diastolic blood pressure of at least 10 mm Hg. Orthostatic changes are calculated as standing – supine.

Baseline values for vital signs will be the observations taken at Visit 2

#### 7.8.4 ECG

Clinically significant findings for ECG will be recorded as baseline conditions or AEs and will be analyzed accordingly.

### **7.8.5** Others

### 24-hour Holter Monitoring

The 24-hour Holter monitoring will be analyzed using descriptive statistics.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8. REFERENCES

- 1 001-MCG-156\_RD-01: "Handling of missing and incomplete AE dates", current version; IDEA for CON.
- 2 *029-DCP-102*: "Noncompartmental Pharmacokinetic Analyses of Clinical Studies", current version; IDEA for CON.
- 3 029-DCG-103: "Noncompartmental Pharmacokinetic Analyses using WinNonlin®", current version; IDEA for CON.
- 4 001-MCG-156: "Handling and summarisation of adverse event data for clinical trial reports and integrated summaries", current version; IDEA for CON.
- 5 *CPMP/ICH/137/95*: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version.
- 6 001-MCG-157: "Display and Analysis of Laboratory Data", current version, IDEA for CON.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 10. HISTORY TABLE

Table 10: 1 History table

This is a revised TSAP including the following modifications to the final TSAP

| Version | Date<br>(DD-Mmm-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Final | 21-Apr-16 | | None | This is the final TSAP without any modification |
| Revised | 08-Aug-17 | | Title page | To indicate that the TSAP covers CTP Amendments 1-3. |
| | | | Section 6.1 | In selected AE tables, HV will be split out to display results for HV_AD and HV_CIAS groups. |
| | | | Section 6.1 | The definition of the start of the baseline period was revised to reflect study conduct differences at the new sites (Subjects at site were inpatients; subjects at sites & were not.) |
| | | | Section 6.2 | CTP Amendment #3 allowed subjects > age 85 to participate in the trial. Exclusion of PK data for subjects outside the original age cut-offs was no longer deemed necessary. The IPV 'Age criteria not met' was removed. |
| | Section 7.8.1 | Section now correctly describes analysis & presentation of AE data based on Version 8 of the guideline. | | |
| | | | Multiple sections | CTP Amendment #1 changed terminology from 'End of Study' to 'End of Trial' for the last study visit. |